CLINICAL TRIAL: NCT00889603
Title: Non-Interventional Study With Aricept® Evess In Patients Diagnosed With Mild And Moderate Alzheimer's Disease Or Vascular Dementia
Brief Title: Non-Interventional Study With Aricept® Evess
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A2501065
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Results first posted 2011-03-31 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer's Disease; Vascular Dementia
Keywords: Aricept® Evess; non-interventional study; Alzheimer's Disease; Vascular Dementia; efficacy; tolerability; safety.
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Aricept® Evess

INTERVENTIONS:
Drug: Aricept® Evess — 5 mg film-coated orodispersible tablets, 10 mg film-coated orodispersible tablets.
  Treatment may be started with 5 mg donepezil/ day (once-a-day dosing) and after four weeks can be titrated to 10 mg/day (once-a-day dosing).

SUMMARY:
The Aricept® Evess study is a prospective, non-comparative, non-interventional study on use of Aricept® Evess in the treatment of out-patients with AD and Vascular Dementia. The 24 week length of the study aims to collect data from a large number of patients (n= 400) on the safety and efficacy at the usual dosage of the product providing an overview of Aricept® Evess profile.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients (male / female), older than 50 years.
* Patients with clinical symptoms of mild and moderate AD and Vascular Dementia.
* MMSE score between 12 - 24.

Exclusion Criteria:

* Patients with a known hypersensitivity to donepezil clorhydrat, piperidine derivatives or any of the excipients of Aricept® Evess.
* Patients with severe impaired hepatic function.
* Patients with pre-existing gastrointestinal ulcer disease.
* Patients with the history of bronchial asthma or chronic obstructive lung disease.
* Patients with the history of serious atrioventricular conduction disturbances.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from those addressing psychiatrists on an outpatient bases, male / female, older than 50 years, being diagnosed with Alzheimer's Disease and Vascular Dementia, with MMSE score between 12 - 24.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Romania (9):
  - Pfizer Investigational Site, Bacau, Jud. Bacau
  - Pfizer Investigational Site, Cluj-Napoca, Jud. Cluj
  - Pfizer Investigational Site, Constanța, Jud. Constanta
  - Pfizer Investigational Site, Craiova, Jud. Dolj
  - Pfizer Investigational Site, Iași, Jud. Iasi
  - Pfizer Investigational Site, Ploieşti, Jud. Prahova
  - Pfizer Investigational Site, Timișoara, Jud. Timis
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Iași

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2501065&StudyName=Non-Interventional%20Study%20With%20Aricept%AE%20Evess%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil: 5 milligrams per day (mg/day), once-a-day dosing and after 4 weeks titrated to 10 mg/day, once-a-day dosing
Period: Overall Study
Arm/Group | Donepezil
Started | 370
Completed | 333
Not Completed | 37
Not completed — Adverse Event | 7
Not completed — Death | 3
Not completed — Lost to Follow-up | 19
Not completed — No longer willing to participant in stud | 4
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil
Number analyzed (Participants) | 370
Age, Customized [Number; unit: Participants]
  Less than 65 years | 71
  65 to 74 years | 130
  75 to 84 years | 142
  Greater than or equal to 85 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 170

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total at Week 24 Last Observation Carried Forward (LOCF)
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranged from 0 - 30, higher score indicated better cognitive state. Change: mean score at Week 24 LOCF minus mean score at baseline.
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of Donepezil and had at least 1 postbaseline efficacy evaluation. LOCF was used. N=number of participants with evaluable data.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 351
Scores on a scale | 1.92 (0.14)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; Mean Difference (Net) = 1.92, 95% CI 2-sided [1.65 to 2.20] — Change from baseline in MMSE at LOCF analyzed using single-sample t-test; a 95% confidence interval (CI) was calculated for mean change at LOCF

2. Secondary Outcome: Change From Baseline in MMSE Total
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranged from 0 - 30, higher score indicated better cognitive state. Change: least squares (LS) mean score at observation minus LS mean score at baseline. Changes from baseline at each week were controlled for baseline MMSE.
Time Frame: Baseline, Week 8, 16, and 24
Population: FAS. N=number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 348
Scores on a scale
  Week 8 (N=348) | 0.92 (0.09)
  Week 16 (N=340) | 1.56 (0.12)
  Week 24 (N=327) | 1.97 (0.14)
Statistical Analysis 1: Comparison: Donepezil; Test type: Superiority or Other; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [0.75 to 1.08] — LS Mean and 95% CI for change from baseline in MMSE Total to Week 8 from repeated-measures mixed model including terms for baseline MMSE and Week
Statistical Analysis 2: Comparison: Donepezil; Test type: Superiority or Other; Mean Difference (Final Values) = 1.56, 95% CI 2-sided [1.32 to 1.80] — LS Mean and 95% CI for change from baseline in MMSE Total to Week 16 from a repeated-measures mixed model including terms for baseline MMSE and Week
Statistical Analysis 3: Comparison: Donepezil; Test type: Superiority or Other; Mean Difference (Final Values) = 1.97, 95% CI 2-sided [1.69 to 2.25] — LS Mean and 95% CI for change from baseline in MMSE Total to Week 24 from a repeated-measures mixed model including terms for baseline MMSE and Week

3. Secondary Outcome: Change From Baseline in Functional Activity Questionnaire (FAQ)
Description: Participants completed the FAQ for physical function. Overall scores could have ranged from 0 (independent) to 30 (dependent) where lower scores represented an improvement in physical function. Change from baseline was to be calculated as baseline scores minus week 24 scores.
Time Frame: Baseline and Week 24
Population: FAS. Data not analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Donepezil
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I) at Week 8
Description: CGI-I: 7-point Investigator-rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement was defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 8
Population: FAS. N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 351
Participants
  Very much improved | 5
  Much improved | 68
  Minimally improved | 194
  No change | 74
  Minimally worse | 8
  Much worse | 2

5. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I) at Week 16
Description: as for outcome 4
Time Frame: Week 16
Population: FAS. N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 341
Participants
  Very much improved | 21
  Much improved | 119
  Minimally improved | 116
  No change | 66
  Minimally worse | 17
  Much worse | 2

6. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I) at Week 24
Description: as for outcome 4
Time Frame: Week 24
Population: FAS. N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 330
Participants
  Very much improved | 33
  Much improved | 129
  Minimally improved | 87
  No change | 62
  Minimally worse | 16
  Much worse | 2
  Very much worse | 1

7. Secondary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I) at Week 24 LOCF
Description: as for outcome 4
Time Frame: Week 24
Population: FAS; LOCF. N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 352
Participants
  Very much improved | 34
  Much improved | 133
  Minimally improved | 95
  No change | 70
  Minimally worse | 17
  Much worse | 2
  Very much worse | 1

8. Secondary Outcome: Number of Participants in Each Patient Domain of Benefit
Description: Participants asked to indicate if the cognition, functionality, and/or behavior domain were most benefited/improved after treatment (dichotomous yes/no endpoints where checking the CRF box next to each domain indicated 'yes' and leaving a box blank indicated 'no').
Time Frame: Week 24
Population: Safety population: all participants who received at least 1 dose of study drug. N=number of participants with evaluable data. Week 24 LOCF not reported as data only collected at Week 24.
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 335
Participants
  Cognition | 202
  Functionality | 215
  Behavior | 193

9. Other Pre Specified Outcome: Number of Participants With Treatment Tolerability
Description: Overall Evaluation of Tolerability at Week 24; 1=Very good, 2=Good, 3=Moderate, 4=Poor
Time Frame: Week 24
Population: Safety population; N=number of particpants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 331
Participants
  Very Good | 186
  Good | 130
  Moderate | 14
  Poor | 1

10. Other Pre Specified Outcome: Number of Participants Receiving Other Medications
Description: Information collected and recorded by investigator in accordance with existing medical records. World Health Organization- Drug (WHO-Drug) coding dictionary applied.
Time Frame: Baseline and Week 24
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Donepezil
Number analyzed (Participants) | 370
Participants
  Baseline | 205
  Week 24 | 270

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a Serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Donepezil
Serious Adverse Events (participants affected / at risk) | 12/370
Other Adverse Events (participants affected / at risk) | 52/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil (N=370)
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Withdrawal syndrome (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil (N=370)
Tinnitus (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 2
Irritability (General disorders) | 1
Weight decreased (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Cerebral disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Neuralgia (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 6
Hypomania (Psychiatric disorders) | 1
Impulse-control disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 13
Restlessness (Psychiatric disorders) | 3
Sleep disorder (Psychiatric disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
FAQ Change from baseline not analyzed, a note to file was issued stating it was removed from protocol but erroneously remained in statistical analysis section. Patient Domain of Benefit, Week 24 LOCF not analyzed; endpoint only collected at Week 24.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.